CLINICAL TRIAL: NCT00519571
Title: Evaluation of the Safety and Efficacy of Using ImplantLock Device - Dental Implant Accessory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Innovative Implant Solutions (Industry)
Responsible Party: Dr. Hanna Levy, Clinical Study Consultant, IIS Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL-01
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Dental Implantation
Keywords: Dental Implantation, Endosseous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: ImplantLock device

INTERVENTIONS:
Device: ImplantLock device — dental implant

SUMMARY:
To investigate the safety and effectiveness of the ImplantLock device and its contribution to 8.0 mm long root-form endosseous implants stability under immediately applied continuous functional loading.

DETAILED DESCRIPTION:
Primary Endpoints

* Serious adverse events occurrence rate (during implantation procedure or following implantation) related to the ImplantLock device will be documented in Serious Adverse Event Form.
* Adverse events occurrence rate (during implantation procedure or following implantation) related to the ImplantLock device will be documented in Adverse Event Form.

Secondary Endpoints

* Determine 8.0 mm long endosseous implant stability while using ImplantLock Device. Stability will be routinely assessed.
* Determine the ability to immediately apply continuous functional loading on 8.0 mm long endosseous implant while using ImplantLock Device. The ability to immediately apply continuous functional loading will be routinely assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female age 18 and up.
* Subject is schedule for endosseous implantation treatment.
* Subject able to comprehend and give informed consent for participation in this study.
* Signed informed consent form.

Exclusion Criteria:

* Subjects suffering from a disease that might disturb bone regeneration healing process e.g. osteoporosis, anemia, etc.
* Acute infection requiring intravenous antibiotics at the time of screening.
* Bleeding disorders.
* Uncontrolled diabetes mellitus
* HIV positive or any other immunosuppressive disorder.
* Renal failure (Serum creatinine >2.0 mg/dl).
* Subject with allergies to metal alloys.
* Coagulation disorder.
* Infection / abscess / pains in treatment target area.
* Pregnant or nursing woman.
* Resent history of alcohol or drug abuse (within the last 2 years).
* Subject is smoking.
* Subject is suffering extreme general weakness.
* Subject objects to the study protocol.
* Known cognitive or psychiatric disorder
* Concurrent participation in any other clinical study.
* Physician objection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events occurrence rate (during implantation procedure or following implantation) related to the ImplantLock device | 12 months

SECONDARY OUTCOMES:
Determine endosseous implant stability while using ImplantLock Device | 12 months
Determine the ability to immediately apply continuous functional loading on endosseous implant while using ImplantLock Device | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Tayeb, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical center, Jerusalem, Israel